CLINICAL TRIAL: NCT01665079
Title: Propofol Effect-Site Target Controlled Infusion in the Obese: Characterization of the Time Profile of Bispectral Index Response.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad del Desarrollo (Other)
Responsible Party: Principal Investigator, Pablo Sepulveda, Profesor Asociado Anestesiología, Universidad del Desarrollo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Propofol TCI obese
Record Dates: First submitted 2012-08-09; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Obesity
Keywords: anaesthetics iv; propofol; pharmacokinetics; pharmacodynamic
MeSH Terms: conditions — Obesity | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Propofol (Experimental): 14 obese patients(IMC>35 kg m-2) scheduled for laparoscopic bariatric surgery
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol was administered by plasma TCI and a bolus dose was given by setting the initial plasma target between 12-16 μg/ml according to the anesthesiologist criteria. The protocol target range was selected based on previous experience using this model in the obese. After the patients reached this target, propofol infusion was stopped until the patients woke up (BIS>75). No other drugs were given during this period. Facemask ventilation was assisted only if necessary to maintain SpO2 > 90%. BIS data and propofol infusion data were automatically recorded every five seconds using the AnestFusor© program. Arterial blood samples of 4 ml for propofol assays were collected at 1, 2, 3, 5, 7 and 10 minutes after the initial bolus dose or until BIS > 75. After the patient woke up the study was considered finished and propofol infusion was restarted according to the anesthesiologist plan.

SUMMARY:
The aim of this study is to characterize the Pharmacokinetic/Pharmacodynamic relationship of a single bolus dose of propofol in obese patients and to extract a time to peak effect (t-peak) from the estimated model parameters.

DETAILED DESCRIPTION:
Target controlled infusion (TCI) is a technique to administer intravenous drugs that allows rapid achievement and maintenance of predetermined drug concentrations, either in plasma (Cp) or at the site of effect (Ce).

To characterize the time profile of propofol effect an additional parameter, the equilibration half time between plasma and effect site (T1/2keo) needs to be incorporated in the pharmacokinetic (PK) model.

ELIGIBILITY:
Inclusion Criteria:

* IMC > 35 kg m-2
* Scheduled for laparoscopic bariatric surgery
* ASA I-II patients
* Between 20 and 60 yr of age.

Exclusion Criteria:

* Patients with allergy to study drugs
* Uncontrolled hypertension
* Heart block greater than first degree
* Take any drug acting in the central nervous system

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Profile of Pharmacokinetic and Pharmacodynamic of an induction bolus dose of propofol in obese patients. | 1, 2, 3, 5, 7 and 10 minutes after the initial bolus dose or until BIS > 75
  Pharmacokinetic parameters (V1, V2, V3, CL, Q)
  Pharmacodynamic parameters (E0, Emax, C50, Gamma, t1/2Ke0, T peak )

CONTACTS AND LOCATIONS:
Overall Officials: Pablo O Sepúlveda, MD, Principal Investigator — Clinica Alemana Universidad del Desarrollo
Locations (1):
- Clinica Alemana, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Derived] Cortinez LI, Sepulveda P, Rolle A, Cottin P, Guerrini A, Anderson BJ. Effect-Site Target-Controlled Infusion in the Obese: Model Derivation and Performance Assessment. Anesth Analg. 2018 Oct;127(4):865-872. doi: 10.1213/ANE.0000000000002814. PMID 29401079